CLINICAL TRIAL: NCT06474676
Title: T Cell Membrane-Anchored Tumor-Targeted IL12 -Modified TIL Cell Therapy (attIL12-TIL) for Advanced/Metastatic Soft Tissue and Bone Sarcoma Patients.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0291; NCI-2024-05385 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Soft-tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A, (Experimental): Participants enrolled in Part A, the dose of attIL2-TIL cell therapy a participant receive will depend on when the participant joins this study. The first group of participants will receive the lowest dose level of attIL2-TIL cell therapy. Each new group will receive a higher dose of attIL2-TIL cell therapy than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of attIL2-TIL cell therapy is found.
  Interventions: Drug: Cyclophosphamide; Drug: T Cell Membrane-Anchored Tumor-Targeted IL12 -Modified TIL Cell Therapy
- Part B (Experimental): Participants enrolled in Part B, will receive attIL2-TIL cell therapy at the recommended dose that was found in Part A.
  Interventions: Drug: Cyclophosphamide; Drug: T Cell Membrane-Anchored Tumor-Targeted IL12 -Modified TIL Cell Therapy

INTERVENTIONS:
Drug: Cyclophosphamide — Given by IV
Drug: T Cell Membrane-Anchored Tumor-Targeted IL12 -Modified TIL Cell Therapy — Given by IV
  Other Names: AttIL2-TIL

SUMMARY:
To find a recommended dose of attIL2-TIL cell therapy that can be given to participant with either relapsed or metastatic sarcomas (has come back or spread to other parts of the body, respectively).

To further test the dose found in Part A to see if it can help to control liposarcoma growth.

DETAILED DESCRIPTION:
Primary Objectives Part A. Determine the safety, maximum tolerated dose and/or recommended phase 2 dose of T cell membrane-anchored tumor- targeted IL12 (attIL12)-TIL cell therapy in combination with cyclophosphamide in participants with advanced/metastatic soft tissue or bone sarcomas Part B. Characterize the safety and tolerability and assess preliminary efficacy of attIL12 TIL cells in combination with cyclophosphamide by evaluating the 4-month progression free survival rate (PFS 4 months) in participants with recurrent unresectable liposarcoma

Secondary Objectives

1) Evaluate the anti-tumor efficacy achieved following adoptive transfer of T cell membrane- anchored tumor- targeted IL12 (attIL12)-TIL cell therapy in combination with cyclophosphamide in participants with advanced/metastatic soft tissue or bone sarcomas

Exploratory Objectives

1. Characterize the immune response following adoptive transfer of attIL12 TIL cell therapy in paired in pre-treatment and on-treatment tumor specimens and peripheral blood samples
2. Assess collagen and FAP changes in pre-treatment and on-treatment tumor specimens and correlate with clinical benefit/anti-tumor response
3. Determine changes in cell surface vimentin (CSV)-positive circulating tumor cells (CTCs) in peripheral blood before and after adoptive transfer of T cell membrane-anchored tumor- targeted IL12 (attIL12)-TIL cell therapy and correlate with clinical benefit/anti-tumor response

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 12 years old
2. Histologically-confirmed locally advanced or metastatic soft tissue or bone sarcoma scheduled to undergo resection or biopsy as part of standard of care
3. Liposarcoma expansion cohort: histologically confirmed unresectable recurrent/metastatic liposarcoma scheduled to undergo resection or biopsy as part of standard of care
4. Participants undergoing resection should have other measurable disease or be high risk for recurrence within 12 month per investigator assessment and has prior approval by PI.
5. Measurable disease according to RECIST 1.1 present prior to infusion of attIL12-TIL. If the only measurable disease is the same as the lesion biopsied for the study, it needs to be at least 2 cm in largest diameter.
6. Participants must have received at least 1 prior line of systemic therapy for the treatment of sarcoma, unless no standard therapy exists for a specific sarcoma subtype.
7. At least 3 weeks must have elapsed since the last cytotoxic chemotherapy or immunotherapy prior to tumor tissue collection. For targeted therapies, at least 4 half-lives or 3 weeks must have elapsed prior to tumor tissue collection (whichever is shorter). Standard of care anti- cancer therapy will be permitted following tumor tissue collection but prior to initiation of cyclophosphamide such that at least 3 weeks must have elapsed since last cytotoxic chemotherapy or immunotherapy prior to starting treatment with cyclophosphamide. For targeted therapies, at least 4 half-lives or 3 weeks must have elapsed prior to initiation of treatment with cyclophosphamide (whichever is shorter). Investigational anti-cancer therapy will not be permitted.
8. At least 2 weeks must have elapsed for palliative radiation to any tumor site other than the tumor site identified for tissue collection
9. Participants must have organ and marrow function as defined below
10. Absolute neutrophil count (ANC) > 1 K/uL, Hemoglobin > 9 g/dL, Platelets > 100 K/mm3
11. Serum creatinine </= 2 mg/dL OR creatinine clearance > 50 mL/min
12. Aspartic transaminase (AST) . 1.5 x upper limit of normal (ULN), Alanine transaminase (ALT) </= 1.5 x ULN, Bilirubin ≤ 1.5 x ULN
13. Women of childbearing potential (WOCBP) must agree to use method(s) of contraception: at least one highly effective or two effective accepted methods of contraception to avoid conception throughout the study in such a manner that the risk of pregnancy is minimized. Suggested precautions should be used to minimize the risk or pregnancy for at least 1 month before start of therapy, and while women are on study for up to 3 months after T cell infusion.

    WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal
14. Men must be willing and able to use an acceptable method of birth control such as latex condom during the dosing period and for at least 3 months after completion of the study agent administration (T cell infusion) if their sexual partners are WOCBP.
15. Signed Informed Consent and if applicable, pediatric assent

Exclusion Criteria:

1. Known sensitivity to cyclophosphamide and/or study agents
2. Active or prior documented autoimmune disease (including inflammatory bowel disease, celiac disease, Wegener syndrome) within the past 2 years. Participants with childhood atopy or asthma, vitiligo, alopecia, Hashimoto syndrome, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded
3. Untreated central nervous system metastatic disease, leptomeningeal disease, or cord compression. Participants previously treated central nervous system metastases that are radiographically and neurologically stable for at least 6 weeks and do not require corticosteroids (of any dose) for symptomatic management for at least 14 days prior to first dose of attIL12-TIL cells are permitted to enroll.
4. Any concurrent chemotherapy, immunotherapy, or biologic or hormonal therapy for cancer treatment at the time of tumor tissue collection or attIL12 TIL cell infusion. Any prior radiation to the tumor site that is being collected for attIL12 TIL production. Palliative radiation to any tumor site within the past 2 weeks. Standard of care anti-cancer therapy will be permitted following tumor tissue collection but prior to initiation of cyclophosphamide as bridging therapy (per section 5.5). Concurrent use of hormones for non-cancer-related conditions (eg, insulin for diabetes and hormone replacement therapy) is acceptable.
5. Unresolved toxicities from prior anticancer therapy, defined as having not resolved to NCI CTCAE v5 Grade 0 or 1 with the exception of alopecia and laboratory values listed per the inclusion criteria. Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by any of the investigational products may be included (eg, hearing loss) after consultation with the PI.
6. History of primary immunodeficiency, solid organ transplantation, or previous clinical diagnosis of tuberculosis.
7. Receipt of live, attenuated vaccine within 28 days prior to the first dose of investigational products.
8. Major surgery (as defined by the investigator) within 4 weeks prior to first dose of treatment. Biopsy as per study protocol is allowed
9. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, unhealed wound, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs from the study agents, or compromise the ability of the participant to give written informed consent. Participants with cognitive impairment, including adults with cognitive impairment such as trisomy 21 or similar conditions are not specifically excluded from participation, such that appropriate written informed consent is obtained from the parent or legal guardian and they are able to complete with the study protocol requirements and treatment.
10. Active concurrent second malignancy
11. Pregnant or lactating women
12. Any positive test result for hepatitis B or C virus indicating acute or chronic infection
13. Known history of testing positive for human immunodeficiency virus or known acquired immunodeficiency syndrome

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Neeta Somaiah, MBBS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org